CLINICAL TRIAL: NCT04562077
Title: Role of Surgery in Treatment of Recurrent Brian Glioma:Prognostic Factors and Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Sayed Mohamad, assistant lecturer, Assiut University
Other Study IDs: surgery in glioma
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Glioma; Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
role of surgery in treatment of recurrent brain glioma prognostic factors and outcome measures Role of surgery : In patients with Grade I gliomas, such as pilocytic astrocytomas, resection is potentially curative.

For more diffuse invasive gliomas (Grade II or higher), initial management typically includes maximal safe resection when possible.

Increasing evidence supports an association between extent of resection and prolonged progression-free and overall survival for patients with diffuse gliomas of all types and grades Many studies reported that more that 90%of patients with glioma showed recurrence at the orginal tumor location.

Review the outcomes of re-operation in treatment of recurrent brain gliomas To determine the prognostic factors which can predict which patient would benefit from multiple surgery .

Trail to Improve the outcome of these patients and decrease rate of complications

ELIGIBILITY:
Inclusion Criteria:

- Patient previously operated and documented as a glioma with clinical and neuroimaging and pathological evidences.

Patients who will undergo re-operation for treatment of a recurrent brain glioma at the time of study(one year) Histological types : Different histological types of glioma.

Exclusion Criteria:

* patients has brain glioma that is de novo patients who are unfit for any neurosurgical interventions. Multicentric recurrent glioma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases that fullfill the selection criteria that will be admitted in the department of neurosurgery Assuit university hospital 01/11/2020 to 30/10/2021.
  Sample size was calculated using Epi- Info7. The previous study reported that, percentage of complications after re-operation in recurrent glioma was 65%. Based on this percentage and with a confidence limits of 10% and a confidence level of 80%, the minimum sample needed for the study was estimated to be 20 patients.
  Patients whose follow-ups will be lost because of death or any other cause will be excluded from this study (expected to be 25%). Additionally, the competence of follow-up will be approved by imaging and medical records.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
karnofsky performance status | 1year
  A standard way of measuring the ability of cancer patients to perform ordinary tasks. The Karnofsky Performance Status scores range from 0 to 100. A higher score means the patient is better able to carry out daily activities. Karnofsky Performance Status may be used to determine a patient's prognosis, to measure changes in a patient's ability to function, or to decide if a patient could be included in a clinical trial. Also called KPS.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed AlGhriany, phD, Study Director — professor of neurosurgery assiut university; Ahmed AlShanawany, phD, Study Director — assistant professor of neurosurgery assiut university; Mohamad S Waer, Principal Investigator — Resident at department of neurosurgery
Locations (1):
- Assuit University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided